CLINICAL TRIAL: NCT02151591
Title: New Approaches to Smoking Cessation in Heavy Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1106008673; K23AA020000-01A1 (NIH)
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Nicotine Dependence; Cigarette Smoking; Alcohol Consumption; Heavy Drinking
Keywords: Quit smoking; Quit drinking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Alcohol Drinking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Counseling for Tobacco and Alcohol (INT) (Experimental): Integrated counseling for smoking and alcohol entails weekly counseling for 12-weeks targeting both behaviors. Participants in this condition will also receive 12 weeks of varenicline (Chantix).
  Interventions: Drug: Varenicline
- Standard Care for Primary Presenting Concern (SC) (Other): Standard care (SC) for primary presenting concern only. For those presenting with the primary concern of tobacco, standard care will involve weekly smoking counseling alone for 12-weeks. For those presenting with the primary concern of alcohol, standard care will involve weekly alcohol counseling alone. Participants in this condition will also receive 12 weeks of varenicline (Chantix).
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — 12-weeks of treatment. Dose will be titrated as follows:
  Days 1-3: 1 0.5mg tablet once per day Days 4-7: 1 0.5mg tablet twice per day Day 8 - Week 11: 1 1mg tablet twice per day
  Other Names: Chantix

SUMMARY:
The purpose of this study is to develop and test an integrated cognitive-behavioral intervention for smoking and alcohol among heavy drinking smokers. The current pre-pilot phase will be used to refine this protocol for the subsequent randomized, controlled pilot phase. The current study phase has two parts: 1) an intake session and brief physical; 2) a 12-week treatment phase in which participants receive varenicline (Chantix) and weekly, personalized counseling.

DETAILED DESCRIPTION:
The purpose of the proposed project is to develop and test a 12-week integrated cognitive-behavioral therapy (CBT) intervention for smoking and alcohol (SA) + varenicline (Chantix) among heavy drinking smokers (i.e., CBT for SA). The project involves two phases. In Phase 1, an open-label pre-pilot study of CBT for SA will be conducted with 10 heavy drinking smokers. The primary results of this phase will be used to refine the CBT for SA protocol. In Phase 2, a randomized, controlled pilot study will be conducted with 40 heavy drinking smokers comparing CBT for SA with standard smoking counseling (SC). All participants in the randomized pilot study will also receive varenicline (Chantix).

Primary and Study Completion dates were changed 6/2016 to reflect an additional year added year to the study.

ELIGIBILITY:
Inclusion Criteria:

1. are at least 18 years of age;
2. report smoking 100 cigarettes over lifetime and currently smoke at least twice weekly on average in the past 90 days and have a urinary cotinine level of >=30ng/mL by semi-quantitative analysis, and/or >= 2 on a NicAlert dipstick
3. are interested in quitting smoking;
4. understand English;
5. exceed National Institute on Alcohol Abuse and Alcoholism heavy drinking criteria (i.e., for men, >14 drinks/week or 5 drinks/day at least once per month over the past 12 months; for women, >7 drinks/week or >4 drinks/day at least once per month over the past 12 months.

Exclusion Criteria:

1. meet criteria for alcohol dependence in the past 12 months that is clinically severe defined by

   * a history of seizures, delirium, or hallucinations during alcohol withdrawal;
   * a Clinical Institute Withdrawal Assessment scale (Sullivan et al., 1989) score of > 8;
   * report drinking to avoid withdrawal symptoms, or d) have had prior treatment of withdrawal;
   * have required medical treatment of alcohol withdrawal within the past 6 months;
2. are currently enrolled in alcohol treatment;
3. meet criteria for drug dependence in the past 12 months; with the exception of marijuana dependence
4. exhibit serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality disorder, organic mood or mental disorders by history or psychological examination;
5. report current suicidality (past 12 months), or report suicide attempts within the past 10 years, assessed with the Columbia Suicide Severity Rating Scale;
6. exhibit current, clinically significant physical disease or abnormality based on medical history, physical examination, or routine laboratory evaluation including:

   * any unexplained elevations in liver enzymes (i.e., transaminases, bilirubin);
   * clinically significant, unstable cardiovascular disease/uncontrolled hypertension;
   * hepatic or renal impairment;
   * severe obstructive pulmonary disease;
   * diabetes mellitus requiring insulin or certain oral medications (i.e., sulfonylureas) and an A1C hemoglobin test score of > 7 for participants not prescribed these medications;
   * baseline systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 95 mm Hg;
7. are cognitively impaired;
8. are unable to read/understand English;
9. are a female of childbearing potential who is pregnant, nursing, or not practicing effective contraception (oral, injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide);
10. report new onset of psychiatric disorders or new psychotropic medications within the past 3 months, except individuals who are on a stable dose of a Selective Serotonin Reuptake Inhibitor for at least two months or who report occasional use of prescription sleep aids that they are willing to discontinue;
11. have used another investigational drug within 30 days or have used medications to treat alcohol (e.g., naltrexone, topiramate, acamprosate, disulfiram) or nicotine use (e.g., clonidine, varenicline, bupropion, nicotine replacement) in the past 3 months or intend to use these medications; (prior use of nicotine replacement in situations where smoking is not permitted (e.g., planes) without the intention to quit smoking is not exclusionary at screening)
12. intend to donate blood or blood products during the treatment phase of the study;
13. have a history of cancer (except treated basal cell or squamous cell carcinoma of the skin);
14. have a history of serious hypersensitivity reactions or skin reactions to varenicline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-reported gender
Enrollment: 26 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available to researchers who request data from the PI
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available upon final publication of the primary paper.
Access Criteria: Upon request to PI

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrated Counseling for Tobacco and Alcohol (INT): Integrated counseling for smoking and alcohol entails weekly counseling for 12-weeks targeting both behaviors. Participants in this condition will also receive 12 weeks of varenicline (Chantix).
  Varenicline: 12-weeks of treatment. Dose will be titrated as follows:
  Days 1-3: 1 0.5mg tablet once per day Days 4-7: 1 0.5mg tablet twice per day Day 8 - Week 11: 1 1mg tablet twice per day
- Standard Care for Primary Presenting Concern (SC): Standard care (SC) for primary presenting concern only. For those presenting with the primary concern of tobacco, standard care will involve weekly smoking counseling alone for 12-weeks. For those presenting with the primary concern of alcohol, standard care will involve weekly alcohol counseling alone. Participants in this condition will also receive 12 weeks of varenicline (Chantix).
  Varenicline: 12-weeks of treatment. Dose will be titrated as follows:
  Days 1-3: 1 0.5mg tablet once per day Days 4-7: 1 0.5mg tablet twice per day Day 8 - Week 11: 1 1mg tablet twice per day
Period: Overall Study
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC)
Started | 13 | 13
Completed | 7 | 10
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: age] | 39.00 (10.59) | 42.62 (13.23) | 40.81 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Abstinence at 6 Months
Description: Number of participants with point prevalence smoking abstinence (i.e., no smoking, not even a puff over the last 7 days) 6 months after treatment completion.
Time Frame: 6 months post treatment start
Population: Number of participants with smoking abstinence at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC)
Number analyzed (Participants) | 13 | 13
Participants | 6 | 3

2. Secondary Outcome: Log Transformed Percentage of Heavy Drinking Days
Description: Log transformed percentage of heavy drinking days 6 months post treatment start.
Time Frame: 6 months post treatment start
Measure: Mean (Standard Error); unit: Mean log transformed percentage score
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC)
Number analyzed (Participants) | 13 | 13
Mean log transformed percentage score | 2.06 (0.40) | 1.45 (0.38)

3. Secondary Outcome: Number of Participants Who Completed Treatment.
Description: To assess feasibility/acceptability, the number of participants who completed treatment will be assessed.
Time Frame: 12 weeks
Population: Number of participants who completed treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC)
Number analyzed (Participants) | 13 | 13
Participants | 7 | 10

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Integrated Counseling for Tobacco and Alcohol (INT) | Standard Care for Primary Presenting Concern (SC)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02151591/Prot_SAP_000.pdf